CLINICAL TRIAL: NCT00925288
Title: Acceptability and Feasibility of a Modified HPV Vaccine Schedule in Brothel Based Female Sex Workers in Peru
Brief Title: Acceptability of Human Papillomavirus (HPV) Vaccine in Female Sex Workers
Acronym: Girasol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); NGO Via Libre (Other); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Neal Halsey, Professor of International Health, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Merck IISP 35706; IRB00001625
Record Dates: First submitted 2009-06-03; First posted 2009-06-22 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Human Papillomavirus Infection
Keywords: Female sex worker; Peru; Cervical infection; Cervical abnormality; Serum antibody; Vaccine acceptance; Alternative schedule; Viral infections; Human papillomavirus vaccine; Human papillomavirus (HPV); non inferiority
MeSH Terms: conditions — Papillomavirus Infections; Virus Diseases | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular schedule (Active Comparator): Duration: Gardasil HPV vaccine administered intramuscularly at 0,2,6 months
  Interventions: Biological: Gardasil
- Modified Schedule (Experimental): Duration: Gardasil HPV vaccine administered intramuscularly at 0,3,6 months
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Gardasil — Dosage Form: 0.5 ml intramuscular injection Dosage: Gardasil 0.5ml suspension Frequency: 3 doses
  Other Names: Human Papillomavirus Quadrivalent Vaccine

SUMMARY:
The primary objectives of this study are to determine the acceptance and potential for the effective use of HPV vaccine in the standard and a modified schedule in female sex workers. Secondary objectives include ascertaining the prevalence of HPV types among female sex workers by age and sexual experience.

DETAILED DESCRIPTION:
FSWs are at higher risk of HPV infection and presumably cervical cancer, and the recently available vaccine has been shown to protect against persistent infection from these types. If this study gives evidence showing the vaccine is acceptable in preventing cervical HPV infection by types 16 and 18 in this population, then the burden of cervical cancer and cancer precursors could be drastically decreased through widespread vaccination of this target group. Vaccination at the point of entry of brothel based sex work may become a requirement to lower the burden of cervical cancer among FSWs and also among all other sex partners of clients of FSWs. A modified schedule may prove beneficial for FSWs in Peru to complete the vaccine regimen.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 and 26 years
* Registered female sex worker living in Lima
* Healthy with no known immune deficiency
* Willing to participate in a study of HPV vaccine including a Pap smear, three pregnancy tests, blood draws, and three vaccine administrations over 7 months
* Willing to provide informed consent

Exclusion Criteria:

* Currently pregnant or planning to get pregnant in the next six months
* Known immune deficiency disorder
* Current receipt of immunosuppressive drugs
* Allergy to yeast or known contraindication to HPV vaccine
* Women who have had their cervix removed
* Previous HPV vaccination
* Current fever over 100 degrees Fahrenheit

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Halsey, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- NGO Via Libre, Lima, Lima Province, Peru

REFERENCES:
- [Background] de Sanjose S, Diaz M, Castellsague X, Clifford G, Bruni L, Munoz N, Bosch FX. Worldwide prevalence and genotype distribution of cervical human papillomavirus DNA in women with normal cytology: a meta-analysis. Lancet Infect Dis. 2007 Jul;7(7):453-9. doi: 10.1016/S1473-3099(07)70158-5. PMID 17597569
- [Background] Mak R, Van Renterghem L, Cuvelier C. Cervical smears and human papillomavirus typing in sex workers. Sex Transm Infect. 2004 Apr;80(2):118-20. doi: 10.1136/sti.2002.003749. PMID 15054172
- [Background] Juarez-Figueroa LA, Wheeler CM, Uribe-Salas FJ, Conde-Glez CJ, Zampilpa-Mejia LG, Garcia-Cisneros S, Hernandez-Avila M. Human papillomavirus: a highly prevalent sexually transmitted disease agent among female sex workers from Mexico City. Sex Transm Dis. 2001 Mar;28(3):125-30. doi: 10.1097/00007435-200103000-00001. PMID 11289192
- [Background] Ford K, Reed BD, Wirawan DN, Muliawan P, Sutarga M, Gregoire L. The Bali STD/AIDS study: human papillomavirus infection among female sex workers. Int J STD AIDS. 2003 Oct;14(10):681-7. doi: 10.1258/095646203322387947. PMID 14596772
- [Background] del Amo J, Gonzalez C, Losana J, Clavo P, Munoz L, Ballesteros J, Garcia-Saiz A, Belza MJ, Ortiz M, Menendez B, del Romero J, Bolumar F. Influence of age and geographical origin in the prevalence of high risk human papillomavirus in migrant female sex workers in Spain. Sex Transm Infect. 2005 Feb;81(1):79-84. doi: 10.1136/sti.2003.008060. PMID 15681729
- [Background] Canadas MP, Bosch FX, Junquera ML, Ejarque M, Font R, Ordonez E, de Sanjose S. Concordance of prevalence of human papillomavirus DNA in anogenital and oral infections in a high-risk population. J Clin Microbiol. 2004 Mar;42(3):1330-2. doi: 10.1128/JCM.42.3.1330-1332.2004. PMID 15004111
- [Background] Kjaer SK, Svare EI, Worm AM, Walboomers JM, Meijer CJ, van den Brule AJ. Human papillomavirus infection in Danish female sex workers. Decreasing prevalence with age despite continuously high sexual activity. Sex Transm Dis. 2000 Sep;27(8):438-45. doi: 10.1097/00007435-200009000-00003. PMID 10987448
- [Background] Tideman RL, Thompson C, Rose B, Gilmour S, Marks C, van Beek I, Berry G, O'Connor C, Mindel A. Cervical human papillomavirus infections in commercial sex workers-risk factors and behaviours. Int J STD AIDS. 2003 Dec;14(12):840-7. doi: 10.1258/095646203322556192. PMID 14678594
- [Background] Anhang R, Goodman A, Goldie SJ. HPV communication: review of existing research and recommendations for patient education. CA Cancer J Clin. 2004 Sep-Oct;54(5):248-59. doi: 10.3322/canjclin.54.5.248. PMID 15371283
- [Background] Roden R, Wu TC. How will HPV vaccines affect cervical cancer? Nat Rev Cancer. 2006 Oct;6(10):753-63. doi: 10.1038/nrc1973. PMID 16990853
- [Background] Burchell AN, Winer RL, de Sanjose S, Franco EL. Chapter 6: Epidemiology and transmission dynamics of genital HPV infection. Vaccine. 2006 Aug 31;24 Suppl 3:S3/52-61. doi: 10.1016/j.vaccine.2006.05.031. Epub 2006 Jun 2. PMID 16950018
- [Background] Stanley M. Immune responses to human papillomavirus. Vaccine. 2006 Mar 30;24 Suppl 1:S16-22. doi: 10.1016/j.vaccine.2005.09.002. PMID 16219398
- [Background] Moscicki AB, Schiffman M, Kjaer S, Villa LL. Chapter 5: Updating the natural history of HPV and anogenital cancer. Vaccine. 2006 Aug 31;24 Suppl 3:S3/42-51. doi: 10.1016/j.vaccine.2006.06.018. Epub 2006 Jun 23. PMID 16950017
- [Background] Holowaty P, Miller AB, Rohan T, To T. Natural history of dysplasia of the uterine cervix. J Natl Cancer Inst. 1999 Feb 3;91(3):252-8. doi: 10.1093/jnci/91.3.252. PMID 10037103
- [Background] Parkin DM, Bray F. Chapter 2: The burden of HPV-related cancers. Vaccine. 2006 Aug 31;24 Suppl 3:S3/11-25. doi: 10.1016/j.vaccine.2006.05.111. PMID 16949997
- [Background] Santos C, Munoz N, Klug S, Almonte M, Guerrero I, Alvarez M, Velarde C, Galdos O, Castillo M, Walboomers J, Meijer C, Caceres E. HPV types and cofactors causing cervical cancer in Peru. Br J Cancer. 2001 Sep 28;85(7):966-71. doi: 10.1054/bjoc.2001.1948. PMID 11592767
- [Background] Clifford GM, Gallus S, Herrero R, Munoz N, Snijders PJ, Vaccarella S, Anh PT, Ferreccio C, Hieu NT, Matos E, Molano M, Rajkumar R, Ronco G, de Sanjose S, Shin HR, Sukvirach S, Thomas JO, Tunsakul S, Meijer CJ, Franceschi S; IARC HPV Prevalence Surveys Study Group. Worldwide distribution of human papillomavirus types in cytologically normal women in the International Agency for Research on Cancer HPV prevalence surveys: a pooled analysis. Lancet. 2005 Sep 17-23;366(9490):991-8. doi: 10.1016/S0140-6736(05)67069-9. PMID 16168781
- [Background] Jacobs MV, Walboomers JM, Snijders PJ, Voorhorst FJ, Verheijen RH, Fransen-Daalmeijer N, Meijer CJ. Distribution of 37 mucosotropic HPV types in women with cytologically normal cervical smears: the age-related patterns for high-risk and low-risk types. Int J Cancer. 2000 Jul 15;87(2):221-7. PMID 10861478
- [Background] Melkert PW, Hopman E, van den Brule AJ, Risse EK, van Diest PJ, Bleker OP, Helmerhorst T, Schipper ME, Meijer CJ, Walboomers JM. Prevalence of HPV in cytomorphologically normal cervical smears, as determined by the polymerase chain reaction, is age-dependent. Int J Cancer. 1993 Apr 1;53(6):919-23. doi: 10.1002/ijc.2910530609. PMID 8386137
- [Background] Kitchener HC, Castle PE, Cox JT. Chapter 7: Achievements and limitations of cervical cytology screening. Vaccine. 2006 Aug 31;24 Suppl 3:S3/63-70. doi: 10.1016/j.vaccine.2006.05.113. PMID 16950019
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Paavonen J, Iversen OE, Olsson SE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, Krogh Gv, Lehtinen M, Malm C, Tamms GM, Giacoletti K, Lupinacci L, Railkar R, Taddeo FJ, Bryan J, Esser MT, Sings HL, Saah AJ, Barr E. High sustained efficacy of a prophylactic quadrivalent human papillomavirus types 6/11/16/18 L1 virus-like particle vaccine through 5 years of follow-up. Br J Cancer. 2006 Dec 4;95(11):1459-66. doi: 10.1038/sj.bjc.6603469. Epub 2006 Nov 21. PMID 17117182
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Halsey NA, Moulton LH, O'Donovan JC, Walcher JR, Thoms ML, Margolis HS, Krause DS. Hepatitis B vaccine administered to children and adolescents at yearly intervals. Pediatrics. 1999 Jun;103(6 Pt 1):1243-7. doi: 10.1542/peds.103.6.1243. PMID 10353936
- [Background] Nunez JT, Delgado M, Giron H, Pino G. Prostitution and other cofactors in preinvasive and invasive lesions of the cervix. Aust N Z J Obstet Gynaecol. 2004 Jun;44(3):239-43. doi: 10.1111/j.1479-828X.2004.00222.x. PMID 15191449
- [Background] Winer RL, Hughes JP, Feng Q, O'Reilly S, Kiviat NB, Holmes KK, Koutsky LA. Condom use and the risk of genital human papillomavirus infection in young women. N Engl J Med. 2006 Jun 22;354(25):2645-54. doi: 10.1056/NEJMoa053284. PMID 16790697
- [Background] Ohshige K, Morio S, Mizushima S, Kitamura K, Tajima K, Suyama A, Usuku S, Tia P, Hor LB, Heng S, Saphonn V, Tochikubo O, Soda K. Behavioural and serological human immunodeficiency virus risk factors among female commercial sex workers in Cambodia. Int J Epidemiol. 2000 Apr;29(2):344-54. doi: 10.1093/ije/29.2.344. PMID 10817135
- [Background] Miller GA, Mendoza W, Krone MR, Meza R, Caceres CF, Coates TJ, Klausner JD. Clients of female sex workers in Lima, Peru: a bridge population for sexually transmitted disease/HIV transmission? Sex Transm Dis. 2004 Jun;31(6):337-42. doi: 10.1097/00007435-200406000-00003. PMID 15167641
- [Background] Trujillo L, Munoz D, Gotuzzo E, Yi A, Watts DM. Sexual practices and prevalence of HIV, HTLV-I/II, and Treponema pallidum among clandestine female sex workers in Lima, Peru. Sex Transm Dis. 1999 Feb;26(2):115-8. doi: 10.1097/00007435-199902000-00010. PMID 10029987
- [Background] Paris M, Gotuzzo E, Goyzueta G, Aramburu J, Caceres CF, Castellano T, Jordan NN, Vermund SH, Hook EW 3rd. Prevalence of gonococcal and chlamydial infections in commercial sex workers in a Peruvian Amazon city. Sex Transm Dis. 1999 Feb;26(2):103-7. doi: 10.1097/00007435-199902000-00008. PMID 10029985
- [Background] Garcia PJ, Chavez S, Feringa B, Chiappe M, Li W, Jansen KU, Carcamo C, Holmes KK. Reproductive tract infections in rural women from the highlands, jungle, and coastal regions of Peru. Bull World Health Organ. 2004 Jul;82(7):483-92. PMID 15508193
- [Background] Sanchez J, Gotuzzo E, Escamilla J, Carrillo C, Phillips IA, Barrios C, Stamm WE, Ashley RL, Kreiss JK, Holmes KK. Gender differences in sexual practices and sexually transmitted infections among adults in Lima, Peru. Am J Public Health. 1996 Aug;86(8):1098-107. doi: 10.2105/ajph.86.8_pt_1.1098. PMID 8712268
- [Background] Sanchez J, Campos PE, Courtois B, Gutierrez L, Carrillo C, Alarcon J, Gotuzzo E, Hughes J, Watts D, Hillier SL, Buchanan K, Holmes KK. Prevention of sexually transmitted diseases (STDs) in female sex workers: prospective evaluation of condom promotion and strengthened STD services. Sex Transm Dis. 2003 Apr;30(4):273-9. doi: 10.1097/00007435-200304000-00001. PMID 12671544
- [Background] Barnabas RV, Laukkanen P, Koskela P, Kontula O, Lehtinen M, Garnett GP. Epidemiology of HPV 16 and cervical cancer in Finland and the potential impact of vaccination: mathematical modelling analyses. PLoS Med. 2006 May;3(5):e138. doi: 10.1371/journal.pmed.0030138. Epub 2006 Apr 4. PMID 16573364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FSWs 18-26 years of age were recruited in person between August 28, 2009 and March 3, 2010 from 49 different sex locales in Lima, Peru by trained medical staff and 8 health promoters. If they fulfilled inclusion criteria, women were asked to report to the study clinic for completion of surveys, vaccination, Pap smears, and counseling.
Pre-assignment Details: Some eligible participants provided a false phone number, did not show up for their study appointment, refused to use birth control when receiving vaccine doses, and reported not having time to participate in the study. After the survey and Pap smear, vaccination was the final step in study enrollment.
Groups:
- Regular Schedule: Duration: 0,2,6 months each dose Dose form: standard injectable HPV4 vaccine Groups: FSWs 18-26 years of age
- Modified Schedule: Duration: 0,3,6 months each dose Dose form: standard injectable HPV4 vaccine Groups: FSWs 18-26 years of age
Period: Overall Study
Arm/Group | Regular Schedule | Modified Schedule
Started | 100 | 100
Completed | 91 | 93
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Regular Schedule: Duration: 0,2,6 months
- Modified Schedule: Duration: 0,3,6 months
- Total: Total of all reporting groups
Arm/Group | Regular Schedule | Modified Schedule | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.86 (2.33) | 22.97 (2.17) | 22.92 (3.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Peru | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Antibody Response to HPV Vaccine for HPV 6,11,16,18.
Description: We measured anitbody response to HPV vaccine for HPV subtypes 6,11,16, and 18. This was compared by study arm, namely the regular and modified vaccination schedules.
Time Frame: Month 7
Population: All participants who returned for the final blood draw considered in the final antibody analysis. The analysis applies to antibody levels after vaccination for HPV6, HPV11, HPV16, and HPV18. This is done for each study arm, namely the regular schedule and the modified schedule.
Measure: Geometric Mean (95% Confidence Interval); unit: Milli Merck Units
Arm/Group | Regular Schedule | Modified Schedule
Number analyzed (Participants) | 89 | 93
Milli Merck Units
  HPV 6 | 1086.49 [854.16 to 1382.0] | 1054.13 [808.42 to 1374.53]
  HPV11 | 745.06 [588.82 to 942.76] | 776.84 [644.03 to 936.21]
  HPV16 | 3235.89 [2661.93 to 3933.61] | 2704.62 [2301.71 to 3178.06]
  HPV18 | 603.39 [487.81 to 746.35] | 531.66 [441.68 to 639.97]
Statistical Analysis 1: Comparison: Regular Schedule vs Modified Schedule; The null hypothesis is that both schedules will provide an equivalent antibody response; Test type: Non-Inferiority or Equivalence — Since the standard schedule is at (0, 2, 6 months), and the modified schedule at (0, 3, 6 months), we will consider this a non-inferiority study. With 80% power, type 1 error of 0.05, standard deviations of 0.6, and an equivalence margin of 0.3, 64 women are needed per group to detect non-inferiority. Having 100 women in each study arm will yield over 94% power to detect non-inferiority of the modified schedule; p > 0.20, Regression, Logistic

2. Primary Outcome: Proportion of Female Sex Workers Who Complete the Three Dose (0, 2, 6 Month) HPV Schedule in a Timely Manner Compared to the Modified (0, 3, 6 Month) Schedule.
Description: Completion of 3 doses of HPV4 vaccine was measured at 6 months for women receiving the vaccine in 0,2,6 month regimen or the modified 0,3,6 month regimen. Completion was measured as receiving dose 3 of the vaccine during the study.
Time Frame: 6 months
Population: All participants were included
Measure: Number; unit: participants
Arm/Group | Regular Schedule | Modified Schedule
Number analyzed (Participants) | 100 | 100
participants | 91 | 93
Statistical Analysis 1: Comparison: Regular Schedule vs Modified Schedule; Completion rates compared in the 2 study arms; Test type: Superiority or Other; p = 0.60, Chi-squared

3. Secondary Outcome: Prevalence of Infection With HPV Subtypes (6,11,16,18) Among Female Sex Workers
Description: Type specific prevalence of HPV6,11,16,18 among study participants, calculated using Linear Array testing.
Time Frame: Baseline
Population: All participants were included in the analysis for baseline HPV DNA prevalence
Measure: Number; unit: participants
Arm/Group | Regular Schedule | Modified Schedule
Number analyzed (Participants) | 99 | 100
participants | 21 | 25
Statistical Analysis 1: Comparison: Regular Schedule vs Modified Schedule; comparison of differences in HPV DNA prevalence by study arm; Test type: Superiority or Other; p = 0.53, Chi-squared

4. Secondary Outcome: Identify Barriers to Acceptance of HPV Vaccine Among Female Sex Workers
Description: Listed doubts about the HPV vaccine. Participants were asked if they had any doubts about the vaccine prior to learning about it from the health professional. Herein we present the total number of participants who reported doubts by study arm.
Time Frame: Month 0
Population: All participants who listed doubts about the vaccine are counted here.
Measure: Number; unit: participants
Groups:
- Regular Schedule: Participants in 0,2,6 month study arm
- Modified Schedule: Participants in 0,3,6 month study arm
Arm/Group | Regular Schedule | Modified Schedule
Number analyzed (Participants) | 100 | 100
participants | 26 | 20

ADVERSE EVENTS:
Arm/Group | Regular Schedule | Modified Schedule
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 0/200 | 0/200

LIMITATIONS AND CAVEATS:
Small time difference between study arms (0,2,6 and 0,3,6 months); We cannot distinguish between antibodies resulting from vaccination and antibodies resulting from natural HPV infection;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No